CLINICAL TRIAL: NCT01112644
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Demonstrate Improvement of Symptoms of RLS in Subjects With Moderate to Severe Idiopathic RLS With Daytime Symptoms Who Take OXN PR Compared to Subjects Taking Placebo (PLA).
Brief Title: Oxycodone/Naloxone Prolonged Release (OXN PR) Compared to Placebo to Demonstrate Improvement in Symptoms of Restless Legs Syndrome (RLS) in Subjects With Moderate to Severe Idiopathic RLS With Daytime Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN3502; 2009-011107-23 (EudraCT Number)
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Moderate to Severe Idiopathic RLS With Daytime Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OXN PR (Experimental): Different daily doses; intake every 12 hours
  Interventions: Drug: Oxycodone naloxone prolonged release tablets (OXN PR)
- PLA (Placebo Comparator): Different daily doses; intake every 12 hours
  Interventions: Drug: Oxycodone naloxone prolonged release tablets (OXN PR); Other: Placebo (PLA)

INTERVENTIONS:
Drug: Oxycodone naloxone prolonged release tablets (OXN PR) — Different daily doses; intake every 12 hours
Other: Placebo (PLA) — Different daily doses; intake every 12 hours
  Arms: PLA

SUMMARY:
The primary objective for the 12-week Titration-/Maintenance Period is:

To demonstrate superior efficacy of OXN PR compared to PLA in the improvement of symptom severity of RLS.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo-controlled, parallel-group, multicenter study to demonstrate improvement of symptoms of RLS in subjects with moderate to severe idiopathic RLS with daytime symptoms who take oxycodone/naloxone prolonged release (OXN PR) compared to subjects taking placebo (PLA).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe idiopathic RLS with daytime symptoms

Exclusion Criteria:

* Females who are pregnant or lactating.
* Subjects with evidence of significant structural abnormalities of the gastrointestinal tract.
* Subjects with evidence of impaired liver/kidney function upon entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in the IRLS score between the two treatment arms will be compared | 12 weeks and a 6 month extension
  The primary objective for the 12-week Titration-/Maintenance Period is:
  IRLS: International Restless Legs Syndrome Study Group Rating Scale Assessment Period baseline (visit 3) to final Maintenance Period.

CONTACTS AND LOCATIONS:
Locations (3):
- Paracelsus Elena Klinik, Kassel, Germany
- Barcelona, Spain
- Gothenburg, Sweden

REFERENCES:
- [Derived] Oertel WH, Hallstrom Y, Saletu-Zyhlarz GM, Hopp M, Bosse B, Trenkwalder C; RELOXYN Study Group. Sleep and Quality of Life Under Prolonged Release Oxycodone/Naloxone for Severe Restless Legs Syndrome: An Analysis of Secondary Efficacy Variables of a Double-Blind, Randomized, Placebo-Controlled Study with an Open-Label Extension. CNS Drugs. 2016 Aug;30(8):749-60. doi: 10.1007/s40263-016-0372-1. PMID 27401882
- [Derived] Trenkwalder C, Benes H, Grote L, Garcia-Borreguero D, Hogl B, Hopp M, Bosse B, Oksche A, Reimer K, Winkelmann J, Allen RP, Kohnen R; RELOXYN Study Group. Prolonged release oxycodone-naloxone for treatment of severe restless legs syndrome after failure of previous treatment: a double-blind, randomised, placebo-controlled trial with an open-label extension. Lancet Neurol. 2013 Dec;12(12):1141-50. doi: 10.1016/S1474-4422(13)70239-4. Epub 2013 Oct 18. PMID 24140442
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN3502